CLINICAL TRIAL: NCT02917031
Title: A 24-Week, Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled Study to Investigate the Effects of Saxagliptin and Sitagliptin in Patients With Type 2 Diabetes Mellitus and Heart Failure
Brief Title: Mechanistic Evaluation of Glucose-lowering Strategies in Patients With Heart Failure
Acronym: MEASURE-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1680C00016
Record Dates: First submitted 2016-09-09; First posted 2016-09-28 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Type 2 Diabetes Mellitus; Heart Failure
Keywords: Type 2 Diabetes Mellitus; Heart Failure; Saxagliptin; Sitagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure | interventions — saxagliptin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Saxagliptin (Active Comparator): one tablet of saxagliptin 5 mg or 2.5 mg + one placebo capsule matching sitagliptin
  Interventions: Drug: Saxagliptin; Drug: Placebo to match sitagliptin
- Sitagliptin (Active Comparator): one capsule of sitagliptin 100 mg or 50 mg + one placebo tablet matching saxagliptin
  Interventions: Drug: Sitagliptin; Drug: Placebo to match saxagliptin
- Placebo (Placebo Comparator): one placebo tablet matching saxagliptin + one placebo capsule matching sitagliptin
  Interventions: Drug: Placebo to match saxagliptin; Drug: Placebo to match sitagliptin

INTERVENTIONS:
Drug: Saxagliptin — 5 mg or 2.5 mg, plain, yellow, biconvex, round, film-coated tablet
  Other Names: Onglyza TM
  Arms: Saxagliptin
Drug: Sitagliptin — 50 mg or 100 mg, gray capsule
  Other Names: Januvia®
  Arms: Sitagliptin
Drug: Placebo to match saxagliptin — 2.5 mg or 5 mg, plain, yellow, biconvex, round, film-coated tablet
  Arms: Placebo; Sitagliptin
Drug: Placebo to match sitagliptin — 50 mg or 100 mg, gray capsule
  Arms: Placebo; Saxagliptin

SUMMARY:
This is a 24 week, multicenter, randomized, double-blind, parallel group, placebo-controlled study to investigate the effects of saxagliptin and sitagliptin on cardiac dimensions and function in patients with type 2 diabetes (T2DM) mellitus and heart failure (HF).

ELIGIBILITY:
INCLUSION CRITERIA:

1. Provision of informed consent prior to any study specific procedure (Pre-screening ICF and Informed Consent collected at screening)
2. Male or female, aged ≥18 years at the time of consent
3. Documented, controlled T2DM, as defined by:

   * Diagnosis of Type 2 DM based on current ADA guidelines (Appendix C) Treatment with stable doses of antidiabetic medications that have not increased or decreased for ≥8 weeks before screening
   * For patients taking insulin, the investigator must query the patient at prescreening or screening regarding his/her usual total daily insulin dose (all types combined) during the previous 8 weeks. Insulin dosages during pre-screening and screening should not vary by more than ±20% on more than two occasions
   * Dosage reductions of insulin and sulfonylurea agents may be considered at randomization to minimize the possibility of hypoglycemia

     * Any reductions in the dosage of insulin and sulfonylurea agents will be at the discretion of the investigator
     * For patients treated with insulin, consider a reduction in dose of 20% at randomization
     * For patients receiving sulfonylurea agents, consider a reduction in dose of 50% or discontinue if on a dosage that is considered low at randomization
4. HFrEF demonstrated by all 3 of the following criteria:

   * History of HF and LVEF ≤45% within the last 6 months (echocardiogram, MRI, left ventriculography, or other accepted methodology). Patients without a recent assessment of LV function will undergo a local echocardiogram at the time of screening to determine ejection fraction
   * Elevated NT-proBNP (>300 pg/mL) during screening
   * Patients should receive background standard of care for HFrEF and be treated according to locally recognized guidelines as appropriate. Guideline-recommended medications should be used at recommended doses unless contraindicated or not tolerated. Therapy should have been individually optimized and stable for >or = 4 weeks (this does not apply to diuretics-see NB below) before screening visit and include (unless contraindicated or not tolerated):
   * an ACE inhibitor, or ARB, or sacubitril/valsartan
   * and
   * a beta-blocker
   * and
   * if considered appropriate by the patient's treating physician; a mineralocorticoid receptor antagonist (MRA)
   * NB: Most patients with heart failure require treatment with a diuretic to control sodium and water retention leading to volume overload. It is recognized that diuretic dosing may be titrated to symptoms, signs, weight, and other information and may thus vary. Each patient should, however, be treated with a diuretic regimen aimed at achieving optimal fluid/volume status for that individual
5. Stable HF, with no evidence of volume overload (no rales, jugular venous distention, peripheral edema) at screening
6. Women of childbearing potential (WOCBP):

   * Must be using appropriate birth control to avoid pregnancy throughout the study and for up to 4 weeks after the last dose of investigational product
   * Must have a negative serum or urine pregnancy test within 72 hours prior to the start of investigational product
   * Must not be breastfeeding.

EXCLUSION CRITERIA:

1. MRI contraindications: all implanted defibrillators; implanted pacemakers and other devices/implants that in the judgment of the investigator preclude an MRI evaluation
2. Patients with atrial fibrillation/flutter, or any rhythm that would impact on MRI imaging quality would be excluded. Patients with a prior history of atrial fibrillation or paroxysmal atrial fibrillation may be eligible for entry into the study based on the investigator's judgment related to the frequency of AF events and the patient's overall condition
3. Body mass index >45 kg/m2 or any condition, including, but not limited to known claustrophobia, that may preclude the ability to perform an MRI scan of acceptable quality, or unwillingness to undergo MRI imaging
4. Receiving incretin therapy (DPP4 inhibitors, GLP-1 mimetics), or having received incretin therapy within the previous 8 weeks of randomization
5. Receiving therapy with a TZD or having received TZD therapy within the previous 8 weeks of randomization
6. Type 1 diabetes mellitus
7. History of unstable or rapidly progressing renal disease
8. A central lab eGFR value <30 mL/min/1.73 m2 on pre-screening or screening
9. New York Heart Association (NYHA) Class IV HF
10. Myocardial infarction, stroke, transient ischemic attack, or coronary revascularization (percutaneous coronary intervention [PCI] or coronary artery bypass graft [CABG]) within the past 3 months of screening
11. Inoperable aortic or mitral valvular heart disease. Recent (within 3 months) or planned valvular heart procedure
12. Heart failure secondary to restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, and hypertrophic obstructive cardiomyopathy
13. Previous cardiac transplantation or transplantation indicated or expected within 6 months of randomization
14. Contraindications to saxagliptin therapy as outlined in the saxagliptin Investigator's Brochure, or to sitagliptin therapy as outlined in the sitagliptin prescribing information
15. Current treatment with strong cytochrome P450 (CYP) 3A4/5 inhibitors
16. Involvement in the planning and/or conduct of the study (applies to both AZ staff and/or staff at the study site)
17. Previous enrollment which disqualifies patient from re-enrollment based on the rules in Section 4.1 of the protocol, or previous randomization in the study
18. Participation in another clinical study with an investigational product during the last 30 days
19. Patients either employed by or immediate relatives of the Sponsor
20. Known human immunodeficiency virus (HIV) infection
21. Severe hepatic disease, including chronic active hepatitis. Positive serologic evidence of current infectious liver disease, including patients who are known to be positive for hepatitis B viral antibody IgM, hepatitis B surface antigen, or hepatitis C virus antibody; or aspartate transaminase (AST) or alanine transaminase (ALT) >3X the upper limit of normal; or total bilirubin (TB) >2 mg/dL
22. Active malignancy requiring treatment at the time of Visit 1(with the exception of successfully treated basal cell or treated squamous cell carcinoma).
23. Pregnant, positive pregnancy test, planning to become pregnant during clinical trial or breast feeding
24. History of any clinically significant disease or disorder which, in the opinion of the investigator, may put the patient at risk because of participation in the study, may influence the results, or may limit the patient's ability to participate in or complete the study
25. Unable or unwilling to provide written informed consent

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (10):
  - Research Site, Torrance, California
  - Research Site, Upland, California
  - Research Site, Miami, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Chicago, Illinois
  - Research Site, The Bronx, New York
  - Research Site, Sayre, Pennsylvania
  - Research Site, Spartanburg, South Carolina
  - Research Site, Houston, Texas
  - Research Site, Milwaukee, Wisconsin
- Research Site, Sofia, Bulgaria
- Research Site, Chicoutimi, Quebec, Canada
- Chile (3):
  - Research Site, Santiago
  - Research Site, Talcahuano
  - Research Site, Viña del Mar
- Hungary (10):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Hajdúszoboszló
  - Research Site, Kecskemét
  - Research Site, Kisvárda
  - Research Site, Nyíregyháza
  - Research Site, Orosháza
  - Research Site, Pécs
  - Research Site, Székesfehérvár
- Romania (2):
  - Research Site, Brasov
  - Research Site, Iași
- Russia (8):
  - Research Site, Izhevsk
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Tomsk
  - Research Site, Yaroslavl
- South Korea (7):
  - Research Site, Busan
  - Research Site, Daejeon
  - Research Site, Gwangju
  - Research Site, Hwaseong-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Wŏnju
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Bangkoknoi
  - Research Site, Chiang Mai
  - Research Site, Khon Kaen
- Ukraine (4):
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Rivne

REFERENCES:
- [Derived] Kanie T, Mizuno A, Takaoka Y, Suzuki T, Yoneoka D, Nishikawa Y, Tam WWS, Morze J, Rynkiewicz A, Xin Y, Wu O, Providencia R, Kwong JS. Dipeptidyl peptidase-4 inhibitors, glucagon-like peptide 1 receptor agonists and sodium-glucose co-transporter-2 inhibitors for people with cardiovascular disease: a network meta-analysis. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD013650. doi: 10.1002/14651858.CD013650.pub2. PMID 34693515
- See also: redacted Protocol (CSP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1680C00016&attachmentIdentifier=40bdcbbf-1c2f-46b3-84aa-09c81798d7ac&fileName=redacted_Protocol_(CSP).pdf&versionIdentifier=
- See also: Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1680C00016&attachmentIdentifier=98837851-1b7e-4675-b9bc-ab19d428b539&fileName=redacted_Statisitical_Analysis_Plan_(SAP).pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met all the inclusion and exclusion criteria were enrolled in 9 countries.
Pre-assignment Details: Participants with documented Ejection Fraction ≤ 45% and NTproBNP > 300 pg/mL had eligibility criteria assessed within 28 days of screening period. Informed consent was obtained prior to any study-related procedures or dosing of IP. 1 subject was excluded from the FAS as incorrectly randomized. This subject was terminated from the study on the day of randomization and no investigational product was dispensed.
Groups:
- Saxagliptin: Participants with an eGFR ≥50 mL/min/1.73m^2 received one saxagliptin 5 mg tablet and one sitaglipitin placebo capsule administered orally once daily for a 24-week treatment period. Participants with an eGFR ≥30 to <50 mL/min/1.73m^2, the dose of saxagliptin was adjusted to one 2.5 mg tablet.
- Sitagliptin: Participants with an eGFR ≥50 mL/min/1.73m^2 received one sitagliptin 100 mg capsule and one saxagliptin placebo tablet administered orally once daily for a 24-week treatment period. Participants with an eGFR ≥30 to <50 mL/min/1.73m^2, the dose of sitagliptin was adjusted to one 50 mg capsule.
- Placebo: Participants recieved one saxagliptin placebo tablet and one sitagliptin placebo capsule administered orally once daily for a 24-week treatment period as a control.
Period: Overall Study
Arm/Group | Saxagliptin | Sitagliptin | Placebo
Started (Participants who received treatment) | 112 | 115 | 120
Completed | 94 | 102 | 105
Not Completed | 18 | 13 | 15
Not completed — Reason not specified | 7 | 5 | 6
Not completed — Development of study-specific withdrawal criteria | 1 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Adverse Event | 4 | 1 | 5
Not completed — Death | 2 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 112 | 115 | 120 | 347
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (7.96) | 64.9 (9.85) | 66.5 (7.84) | 65.4 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 37 | 108
  Male | 77 | 79 | 83 | 239
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 16 | 17 | 43
  Not Hispanic or Latino | 102 | 99 | 103 | 304
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 17 | 17 | 15 | 49
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 4
  White | 94 | 98 | 102 | 294
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Left Ventricular End Diastolic Volume (LVEDV) Index Measured by Magnetic Resonance Imaging (MRI) at 24 Weeks
Description: MRI was performed to evaluate LVEDV at baseline and Visit 10 (Week 24). Evaluated to exclude an increase in left ventricular end diastolic volume (LVEDV) index of greater than 10% of the overall baseline value (noninferiority margin) in patients with T2DM and HF treated with saxagliptin for 24 weeks, compared to placebo. Baseline is last assessment on or before the date of first dose.
Time Frame: Baseline to 24 weeks
Population: Full analysis set (FAS): All randomised patients who took at least one dose of the study medication. Here, overall number of participants analyzed presents only those participants who were analyzed for this particular outcome measure.
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 96 | 106
mL/m^2 | -3.395 (15.3412) | -0.716 (18.1178)
Statistical Analysis 1: Comparison: Saxagliptin vs Placebo; Change from baseline, saxagliptin versus placebo; Test type: Superiority; p = 0.252, ANCOVA; Mean Difference (Final Values) = -2.595, 95% CI 2-sided [-7.040 to 1.850]

2. Secondary Outcome: Change From Baseline in Left Ventricular End Systolic Volume (LVESV) Index, Measured by MRI at 24 Weeks.
Description: Evaluation of the effects of saxagliptin compared to placebo on left ventricular end systolic volume (LVESV) index, after 24 weeks in patients with T2DM and HF.
Time Frame: Baseline to week 24
Population: FAS: All randomised patients who took at least one dose of the study medication. Here, overall number of participants analysed presents only those participants who were analyzed for this particular outcome measure.
Measure: Mean (Standard Deviation); unit: mL/m2
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 96 | 106
mL/m2 | -2.555 (12.4136) | -0.839 (17.2458)
Statistical Analysis 1: Comparison: Saxagliptin vs Placebo; Saxagliptin: Change from baseline; Test type: Superiority; p = 0.425, ANCOVA; Mean Difference (Final Values) = -1.631, 95% CI 2-sided [-5.635 to 2.373]

3. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) Measured by MRI at 24 Weeks.
Description: Evaluation the effects of saxagliptin compared to placebo on left ventricular end systolic volume (LVESV) index, left ventricular ejection fraction (LVEF), and left ventricular mass (LVM) after 24 weeks in patients with T2DM and HF.
Time Frame: Baseline to week 24
Population: Full analysis set (FAS): All randomised patients who took at least one dose of the study medication. Here, overall number of participants analysed presents only those participants who were analyzed for this particular outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 96 | 106
Percentage | 0.533 (7.1971) | 0.298 (7.2843)
Statistical Analysis 1: Comparison: Saxagliptin vs Placebo; Saxagliptin vs Placebo: Change from baseline; Test type: Superiority; p = 0.925, ANCOVA; Mean Difference (Final Values) = 0.100, 95% CI 2-sided [-1.996 to 2.197]

4. Secondary Outcome: Change From Baseline in Left Ventricular Mass (LVM) Measured by MRI at 24 Weeks.
Description: Evaluation of the effects of saxagliptin compared to placebo on left ventricular mass (LVM) after 24 weeks in patients with T2DM and HF.
Time Frame: At 24 week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Gram
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 96 | 106
Gram | -4.211 (16.6003) | -0.758 (16.1763)
Statistical Analysis 1: Comparison: Saxagliptin vs Placebo; Saxagliptin vs placebo: Change from baseline; Test type: Superiority; p = 0.105, ANCOVA; Mean Difference (Final Values) = -3.605, 95% CI 2-sided [-7.970 to 0.760]

5. Secondary Outcome: Change From Baseline in NT-proBNP After 24 Weeks of Treatment
Description: Evaluation of the effects of saxagliptin compared to placebo on N-terminal prohormone of brain natriuretic peptide (NT-proBNP) after 24 weeks of treatment.
Time Frame: Baseline to Week 28 (End of Study visit [EoS])
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 93 | 104
pg/mL | -277.525 (1324.7471) | -61.895 (3415.9525)
Statistical Analysis 1: Comparison: Saxagliptin vs Placebo; Saxagliptin vs placebo: Change from baseline; Test type: Superiority; p = 0.796, ANCOVA; Ratio for relative change = 0.971, 95% CI 2-sided [0.777 to 1.214]

6. Secondary Outcome: Number of Participants With Adverse Events
Description: Assessment of safety and tolerability of saxagliptin and sitagliptin treatment in patients with T2DM and HF
Time Frame: From screening (Days -28 to -1) until Week 28 (follow-up visit)
Population: Safety analysis set (SAS): All randomised patients who took at least one dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Saxagliptin | Sitagliptin | Placebo
Number analyzed (Participants) | 112 | 115 | 120
Participants
  Any AE | 53 | 51 | 58
  Any severe AE | 9 | 13 | 14
  Any treatment related AE | 3 | 4 | 0
  Any AE with outcome Death | 2 | 3 | 4
  Any SAE | 17 | 19 | 29
  Any treatment related SAE | 0 | 0 | 0
  Any SAE leading to discontinuation of study treatment | 1 | 0 | 4
  Any AE leading to discontinuation of study treatment | 5 | 3 | 7
  Any Adverse event of special interest | 12 | 15 | 16

ADVERSE EVENTS:
Time Frame: From screening (Days -28 to -1) until Week 28 (follow-up visit)
Description: An AEs is the development of an undesirable medical condition or the deterioration of a preexisting medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product.
Arm/Group | Saxagliptin | Sitagliptin | Placebo
All-Cause Mortality (participants affected / at risk) | 2/112 | 3/115 | 4/120
Serious Adverse Events (participants affected / at risk) | 17/112 | 19/115 | 29/120
Other Adverse Events (participants affected / at risk) | 8/112 | 9/115 | 8/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin (N=112) | Sitagliptin (N=115) | Placebo (N=120)
Cardiac failure (Cardiac disorders) | 7 | 5 | 6
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 1
Acute hepatitis B (Infections and infestations) | 0 | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1 | 2
Cardiac death (General disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Back disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saxagliptin (N=112) | Sitagliptin (N=115) | Placebo (N=120)
Cardiac failure (Cardiac disorders) | 2 (2) | 5 (5) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT02917031/Prot_002.pdf
  • Statistical Analysis Plan (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT02917031/SAP_001.pdf